CLINICAL TRIAL: NCT01574495
Title: Evaluating Error Augmentation for Neurorehabilitation
Acronym: VREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Patton, Co-Director, Robotics Laboratory, Sensory Motor Performance Program, Rehabilitation Institute of Chicago, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H133E0700 13; STU00002311 (Other: NU IRB)
Record Dates: First submitted 2012-02-28; First posted 2012-04-10 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Stroke
Keywords: stroke; error augmentation; arm recovery; massed practice
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Error Augmentation-Control (Experimental)
  Interventions: Other: Error Augmentation
- Control-Error Augmentation (Experimental)
  Interventions: Other: Error Augmentation

INTERVENTIONS:
Other: Error Augmentation — error augmentation for arm motor recovery in individuals with stroke
  Other Names: Error Augmentation-Control; Control-Error Augmentation

SUMMARY:
This is a sub-project of a larger NIDRR Grant. One promising form of robotic training that leverages the power of neuro-plasticity is error augmentation. In this paradigm the computer singles out and magnifies a stroke survivor's movement errors from a desired trajectory, thus forcing the subjects to strengthen their control. Using the VRROOM, a state-of-the-art system which uses haptics (robotic forces) and graphics (visual display) interfaces, a subject's desired trajectory can be determined and the movement errors can be amplified in real-time with dramatic results. This project evaluates a practical approach of error augmentation, using therapist-driven trajectories. The investigators intend to determine clinical efficacy of several types of therapist-assisted error augmentation on retraining the nervous system in functional activities. The investigators will test two experimental treatments in a crossover design. The investigators hypothesize that combined haptic and visual error augmentation will lead to the best functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* adult (age >18)
* survived a single cortical stroke at least 6 months previously involving ischemia or hemorrhage of the middle cerebral artery (MCA),
* demonstrated the presence of some active shoulder and elbow movement (characterized by Fugl-Meyer Assessment Upper Extremity scores ranging from 15-50 for ARM 1; 25-50 for ARM 2).

Exclusion Criteria:

* diffuse or multiple lesion sites or multiple stroke events
* bilateral paresis
* severe spasticity or contracture (Modified Ashworth ≥3
* severe concurrent medical problems
* severe sensory deficits
* cerebellar strokes resulting in severe ataxia
* significant shoulder pain
* focal tone management with Botulinim Toxin (Botox®) injection to the hemiparetic upper extremity (UE) within the previous four months,
* aphasia that would influence the ability to perform the experiment
* cognitive impairment (Mini Mental State Examination < 23/30)
* affective dysfunction that would influence the ability to perform the experiment
* depth perception impairment (< 3 on Stereo Circle Test)
* visual field cut or hemispatial neglect that would influence the ability to participate in the activity
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Arm motor recovery scores on the Fugl-Meyer | Change from baseline in Fugl-Meyer to 11 weeks (with assessment periods occurring at 2 weeks, 3 weeks, 4 weeks, 6 weeks, 7 weeks, and 11 weeks for ARM 1; at start of week 1 (pre-eval), end of week 2 (post), and end of week 3 (1 week follow-up) for ARM 2)
  Change from baseline in arm motor recovery as measured by Fugl-Meyer

SECONDARY OUTCOMES:
Number of blocks transferred in Box and Blocks Test | same as primary
  Change from baseline in number of blocks transferred during Box and Blocks Test
Time and Quality of movement scores on the Wolf Motor Function Test | same as primary
  Change from baseline in arm motor recovery as measured by time scores and ability scores on the Wolf Motor Function test
Time scores and Ability scores on the Assessment of Simple Functional Reach Test | same as primary (not used for ARM 2)
  Change from baseline in arm motor recovery as measured by time scores and ability scores on the Assessment of Simple Functional Reach Test
Quantity and Quality with Motor Activity Log | same as primary but added for ARM 2
  Change in baseline of self-reported quantity and quality of functional movements utilizing involved extremity

CONTACTS AND LOCATIONS:
Overall Officials: James Patton, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States